CLINICAL TRIAL: NCT00446628
Title: Pittsburgh Influenza Prevention Project
Brief Title: Project to Investigate Ways to Reduce the Spread of Influenza in Schools and Households With Children
Acronym: PIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kiren Mitruka (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kiren Mitruka, Medical officer, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCPDCID-CC-0612047; CDC-U01 CI000435-01 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
Keywords: Non-pharmaceutical; influenza; pandemic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): Five elementary school received intervention consistin of training in hand and respiratory hygiene, and access to hand sanitizer
  Interventions: Behavioral: behaviors reducing spread of influenza
- control (No Intervention): Five elementary school received no training or hand sanitizer.

INTERVENTIONS:
Behavioral: behaviors reducing spread of influenza — Non-pharmaceutical interventions for flu prevention
  Arms: intervention

SUMMARY:
The purpose of this study is to understand the spread of influenza (flu) in schools and households with elementary (K-5) school children, and develop ways to reduce the flu using non-pharmaceutical means.

DETAILED DESCRIPTION:
Pandemic influenza threatens to cause substantial disability, death, and societal disruption and to overwhelm health care systems in the United States and around the world. Because effective vaccines may not be available during the initial months of a pandemic, and because anti-viral medication is both largely ineffective and in short supply, non-pharmacological personal protection and behavioral changes may be the only means to combat the epidemic. In our computational modeling work (through the Models of Infectious Disease Agent Study network), we have shown the potential value of multiple targeted and layered non-pharmacological interventions in blunting the peak impact and slowing of a pandemic (Nature, in press).

Phase 1 of the project will be a pilot study in two elementary schools in the City of Pittsburgh. The project has already obtained agreement to collaborate from the Pittsburgh Public School System and we have assembled a multi-disciplinary team of epidemiologists, systems analysts, modelers, community and minority health workers, and virologists to implement the project. Phase one was in 2 schools.

Phase 2 will be similar to Phase 1 with the addition of additional schools and application of a "hygiene" intervention to selected schools and families. Phase 2 is in 10 schools with 3800 students.

Specific aims (year 02):

Primary

1. Measure the effectiveness of non-pharmaceutical interventions (NPIs) in reducing influenza rates among enrolled students in the intervention and control schools when influenza is known to be circulating in the community. [Note: Enrolled, for purposes of PIPP, will indicate students who present with ILI, consent to participate, and are tested for influenza during the flu season.] Secondary: School-Based
2. Measure number of absentees and determine the reason for absence by using a school based absentee illness surveillance system prior to and through the end of influenza season.
3. Measure the effectiveness of NPIs in reducing absenteeism from all causes, including illness/URI, illness/ILI, illness/other, and illness/GI through the end of influenza season.
4. Measure the effectiveness of NPIs in reducing secondary spread of ILI within classrooms of participating schools.
5. Assess adoption of NPI behaviors and activities in classrooms of intervention schools.

   Secondary: Home-Based
6. Measure the effectiveness of NPIs in reducing secondary cases of ILI within families of enrolled school children with influenza.
7. Assess adherence of families of enrolled school children with influenza to isolation-related NPI behaviors and activities.

   Tertiary
8. Measure correlation between rapid flu testing and PCR testing for influenza.
9. Collect and archive influenza specimens for future molecular epidemiological studies.
10. Contribute a sample of influenza-positive specimens to the CDC for national influenza surveillance purposes.

ELIGIBILITY:
Inclusion Criteria (student):

* Students in grades K-8 with a current influenza-like illness (ILI) during flu season.ILI defined as an oral or aural temperature > 100 °F AND either new onset cough or sore throat.Flu season is defined as December, 2006 through March/April, 2007.
* Parental consent and student assent.

Inclusion Criteria (household members):

* Shares living space with K-8 child who has current influenza infection.
* Parental consent and child assent in the case of minors.
* Individual consent if over the age of 18.
* Will continue in the study even if student with confirmed influenza withdraws from the study.

Exclusion Criteria (student):

* The participant has a medical or mental health condition which in the judgment of the investigator is a barrier to safe participation.
* The participant is unable to tolerate a swab or capillary finger stick.
* There is a delay in notification or testing such that symptoms have resolved.

Exclusion Criteria (household):

* The participant has a medical or mental health condition which in the judgment of the investigator is a barrier to safe participation.
* The participant is younger than 6 months.
* The participant is unable to tolerate a swab or capillary finger stick.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3360 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Burke, MD, Principal Investigator — University of Pittsburgh; Sam Stebbins, MD, MPH, Principal Investigator — University of Pittsburgh School of Public Health
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No